CLINICAL TRIAL: NCT02071030
Title: The Efficacy of Cone Beam Computed Tomography (CBCT) Compared to Panoramic Radiography Prior to Third Molar Removal; a Multicentre Randomised Controlled Trial
Brief Title: The Efficacy of Cone Beam Computed Tomography (CBCT) Compared to Panoramic Radiography Prior to Third Molar Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL nr.: 40492.091.12
Record Dates: First submitted 2014-02-11; First posted 2014-02-25 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Inferior Alveolar Nerve Injury
Keywords: CBCT; Third molar removal; Inferior alveolar nerve injury

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- CBCT (Other): Cone Beam CT
  Interventions: Procedure: Third molar removal
- Panoramic radiograph (Other)
  Interventions: Procedure: Third molar removal

INTERVENTIONS:
Procedure: Third molar removal — Surgically removing the third molar in the lower jaw

SUMMARY:
The purpose of this study is to evaluate the efficacy and cost-effectiveness of Cone Beam Computed Tomography (CBCT) compared to panoramic radiography prior to removal of third molars in reducing patient's morbidity. Adults having a close relationship between the mandibular canal and one or both lower third molars, as diagnosed from digital panoramic radiographs will be recruited for this randomised controlled trial. In one trial arm, patients will receive the standard digital panoramic radiograph prior to third molar surgery. In the second arm, subjects will undergo an additional Cone Beam Computed Tomography (CBCT) prior to third molar surgery.

All patients require a postoperative visit one week after surgery to assess the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 year
* mandibular canal is superimposed more than one half by the roots of the third molar as assessed on panoramic radiograph.

Exclusion Criteria:

* pregnancy
* radiological evidence of cyst an tumors
* indication for removal under general anesthesia
* preoperative neurosensory alterations
* existence of an external CBCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with inferior alveolar nerve (IAN) injury | 1 week after surgery

SECONDARY OUTCOMES:
Change in Oral Health related quality of life score | 1 week after surgery

OTHER OUTCOMES:
Costs of imaging, treatment and day's of work. | 2 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Centre. Department of Oral & Maxillofacial Surgery, Nijmegen, Netherlands

REFERENCES:
- [Derived] Ghaeminia H, Gerlach NL, Hoppenreijs TJ, Kicken M, Dings JP, Borstlap WA, de Haan T, Berge SJ, Meijer GJ, Maal TJ. Clinical relevance of cone beam computed tomography in mandibular third molar removal: A multicentre, randomised, controlled trial. J Craniomaxillofac Surg. 2015 Dec;43(10):2158-67. doi: 10.1016/j.jcms.2015.10.009. Epub 2015 Oct 23. PMID 26596360